CLINICAL TRIAL: NCT04658732
Title: A Comparative Study of Oral Gabapentin, Oral Alprazolam and Intravenous Dexmedetomidine on Perioperative Anxiety and Pain During Posterior Segment Eye Surgery Under Peribulbar Block : a Randomized, Double-blind Study.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ehab Tarek Fahmy (Other)
Responsible Party: Sponsor-Investigator, Ehab Tarek Fahmy, MSc, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-240-2019
Record Dates: First submitted 2020-12-05; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Sedation for Patients Undergoing Peribulbar Block
MeSH Terms: interventions — Gabapentin; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Randomized double blinded study.
Who Masked: Participant, Care Provider
Masking Description: Patients will be randomly allocated by a computer-generated table into one of the study groups; the randomization sequence will be concealed in sealed opaque envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alprazolam (A group) (Experimental): patients in this group will receive 0.25 mg Alprazolam (2 tablets of Xanax 0.125 mg manufactured by Pfizer.
  Interventions: Drug: Administration of Alprazolam , Gabapentin , Dexmedetomidine
- Gabapentin (G group) (Experimental): patients in this group will receive 600mg Gabapentin (2 capsules of Neurontin 300 mg manufactured by Pfizer.
  Interventions: Drug: Administration of Alprazolam , Gabapentin , Dexmedetomidine
- Dexmedetomidine (D group) (Experimental): Dexmedetomidine 0.25 µg/kg loading dose will be infused intravenously over 10 minutes through syringe pump before surgery in the control group (Prepared using Precedex vial 200mcg/2ml manufactured by Hospira Inc, Highway 301,Rocky Mount,NC 278001 USA)
  Interventions: Drug: Administration of Alprazolam , Gabapentin , Dexmedetomidine

INTERVENTIONS:
Drug: Administration of Alprazolam , Gabapentin , Dexmedetomidine — Patients will be allocated into one of the 3 groups: Alprazolam (A group), Gabapentin (G group) and Dexmedetomidine (D group) as control group. Alprazolam group (n=15): patients in this group will receive 0.25 mg Alprazolam (2 tablets of Xanax 0.125 mg manufactured by Pfizer). Gabapentin group (n=15): patients in this group will receive 600mg Gabapentin (2 capsules of Neurontin 300 mg manufactured by Pfizer).Control group (n=15): patients in this group will receive 2 tablets of multivitamin (Vitamax manufactured by GlaxoSmithKline S.A.E) as placebo to ensure blindness of the study. The study drug will be received 120 minutes before the operation.

SUMMARY:
We hypothesized that gabapentin when given orally as a premedication in patients who perform posterior segment eye surgery under peribulbar block would provide adequate anxiolysis and arousable sedation as alprazolam and dexmedetomidine with minimal side effects .

DETAILED DESCRIPTION:
The principle goal of sedation for eye surgery is to prepare the patients to stay calm during surgery. Both insufficient sedation and deep sedation may lead to sudden movements by patients, which may potentially result in harmful complications during eye surgery. Several drugs such as propofol, opioids, and dexmedetomidine have been used for sedation during this procedure [1]. However, each of these drugs has its own limitations, leading to impairment of patient's cooperation during surgery. Therefore, the potential clinical advantages of newly-marketed therapeutic drugs should be thoroughly evaluated. [2] Benzodiazepines are amongst the most popular preoperative medication to produce anxiolysis, amnesia, and sedation for the patients coming for surgery [3]. Benzodiazepines are reported to be paradoxically associated with the increased episodes of arousal during sleep, restlessness, and hangover effects [4]. Alprazolam, a benzodiazepine class of antipsychotic drugs, is more anxioselective than the other premedicants of this group like midazolam, lorazepam, or diazepam [5]. It has also been reported to show arousal episodes and may cause psychomotor impairment which is a disadvantage to be used in elderly in general and in day case in particular [4,6].

Gabapentin is well-tolerated drug that is associated with anxiolytic and antinociceptive properties [2]. It is reported that gabapentin has anxiolytic [7] and antinociceptive effects [8,9]. In another study, it is claimed that this drug does not depress respiration with no effect on gastric mucosa, platelets, and renal function [9]. Moreover, gabapentin seems to be an anxiolytic without amnesic effects which is an important advantage for elderly patients. Leung and colleagues reported that delirium is significantly less in patients receiving gabapentin before spine surgery[10].

Dexmedetomidine, a highly selective α2 agonist, has been widely used as a sedative in a variety of clinical settings owing to its analgesic properties, minimal respiratory depression and easy arousability [11,12].Hypotension and bradycardia, the most frequent side effects of dexmedetomidine [12], occur in a dose-related manner [13,14]. To avoid these side effects, a dose adjustment is required. For procedural sedation, a loading dose of 0.25μg/kg over 10 min followed by maintenance dose of 0.25μg/kg/h provides an adequate level of sedation, stable hemodynamics and better surgeon satisfaction [15].

In this study, we planned to compare the sedative effects of oral gabapentin, alprazolam and intravenous of dexmedetomidine on various parameters including anxiety, sedation and orientation. In our literature review, we could not find any study comparing the effect of gabapentin and alprazolam on anxiety, pain, sedation scores, satisfaction of surgeon, and hemodynamic parameters in posterior segment eye surgery under peribulbar block.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 45 to 65 years old, of both sexes.
* ASA 1-2.
* Undergo posterior eye surgery (vitrectomy and retinal detachment) under peribulbar block.

Exclusion Criteria:• Patient refusal.

* Uncooperative patient.
* Communication difficulty resulting from deafness or language barrier.
* Chronic use of narcotics, barbiturate, psychotropic medications or claustrophobia.
* Body weight less than 40 kg or more than 100 kg.
* Known allergy to local anesthetics or any of the study drugs.
* ASA 3-4.
* Inability to lie supine for the time of surgery or involuntary movement.
* Patients with baseline heart rate (HR) <60/min, severe left ventricular dysfunction (EF <30%), hypovolaemia with systolic blood pressure (SBP) <90 mmHg, Mobitz type 2 or 3rd degree heart block, severe valvular disease (valve stenosis/regurgitation), asthma, chronic cough, upper respiratory tract infection within the previous 2 weeks, chronic renal failure and hepatic impairment will be excluded from the study.
* Patients on medications can affect the removal of alprazolam from the body, which may affect how alprazolam works. Examples include azole antifungals (such as itraconazole, ketoconazole),cimetidine, certain antidepressants (such as fluoxetine, fluvoxamine, nefazodone ),drugs to treat HIV( delavirdine, protease inhibitors such as indinavir), macrolide antibiotics (such as erythromycin), rifamycins (such as rifabutin), St.John's Wort and drugs used to treat seizures (such as phenytoin).
* Patients with myasthenia gravis or myoclonus problems.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
primary outcome | intraoperative and 2 hours postoperative . along time of the study
  The sedation level of patients using Ramsay sedation scale (RSS) [19] during surgery will be assessed every 5 min for the first 15 min (5, 10, 15), every 15 min until the end of surgery and every 30 min for 2 h in the post-operative ward.

SECONDARY OUTCOMES:
Secondary outcome | intraoperative and 2 hours postoperative . along time of the study
  • The verbal pain score (VPS) ranging from 0 to10 (0 = no pain and 10 = worst pain imaginable) will be fully explained to patients

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy School of Medicine, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided